CLINICAL TRIAL: NCT05784857
Title: The Effect of Touch Methods on Pain and Physiological Parameters in Preterm Infants During Endotracheal Aspiration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2022/17
Record Dates: First submitted 2023-02-28; First posted 2023-03-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Preterm; Pain; Infant ALL
Keywords: touch; preterm infant; pain
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- No Intervention and Touch Group (Other): Each intubated infant will be follewed up during 3 aspiration procedures. Different touching techniques will be used for preterm infants in each aspiration application.
  The first aspiration procedure will be performed without intervention. During the second aspiration procedure, yakson touch will be applied.Third aspiration procedure, gentle human touch will be applied.
  Interventions: Other: Touch Methods

INTERVENTIONS:
Other: Touch Methods — The Yakson touch method continue for 15 minutes with steady touch (5 minutes), compassionate caressing (5 minutes), and repetition of steady touch (5 minutes). In this method, the palms of the practitioner and all fingers keep in close contact so that the babies don't feel pressure.
  Gentle human touch refers to steady contact of the skin without caressing or massaging. While the practitioner place one hand on the crown of the preterm infant on the eyebrow line with the fingertip touch for 15 minutes, the other hand was place on the lower abdomen covering the waist and hip of the infants.

SUMMARY:
Recurrent and painful interventions such as heel lancing, venipuncture, dressing change, endotracheal aspiration are frequently performed in neonatal intensive care units (NICU). Touch is one of the infant's earliest developing senses. Therefore it is very important among individualized supportive care practices. Correct stimulation of the infant's sense of touch affects psychosocial development positively. In addition, it is reported that touch has a calming and analgesic effect during invasive interventions. Therefore, there is a need for touch appropriate for development of newborn.

The aim of this study was determine the effect of Yakson and Gentle Human Touch on pain and physiologic parameters in preterm infants during endotracheal aspiration.

DETAILED DESCRIPTION:
It was designed as a prospective, quasi-experimental.In this study, each intubated infant will be followed up during 3 aspiration procedures. The first aspiration procedure will be performed without intervention. During the second and third aspiration procedure, yakson and gentle touch will be applied, respectively.Physiological parameters and pain score of newborn will be evaluated before, during and immediately after aspiration.

Yakson touch: Yakson touch is defined in traditional Korean culture as a kind of therapeutic touch that a mother believes will treat her sick child by stroking it with a compassionate, sincere and loving attitude. The Yakson protocol was developed by Im and Kim (2009) in an understandable form that can be easily implemented. While newborn is in supine position, practitioner applies Yakson touch. The Yakson touch method continue for 15 minutes with steady touch (5 minutes), compassionate caressing (5 minutes), and repetition of steady touch (5 minutes). In this method, the palms of the practitioner and all fingers keep in close contact so that the babies don't feel pressure.

1. Steady touch (5 minutes): One hand rest on the chest and abdomen of the preterm infant, while the other hand support the back and hip of the preterm infant.
2. Compassionate Caress (5 minutes): In the same hand position, the practitioner repeat caressing and resting for 5 minutes: Caress (1 minutes), rest (30 seconds), caress (1 minutes), rest (30 seconds), and caress (2 minutes). The practitioner caress the infants' chest and belly with a 1 cm diameter clockwise circular movement every 10 second.
3. Steady touch (5 minutes): The practitioner follow the steady touch procedure as previously describe.

Gentle Human Touch: Gentle human touch refers to steady contact of the skin without caressing or massaging. While the practitioner place one hand on the crown of the preterm infant on the eyebrow line with the fingertip touch for 15 minutes, the other hand was place on the lower abdomen covering the waist and hip of the infants.

ELIGIBILITY:
Inclusion Criteria:

* The gestational week of the infant is less than 38
* Absence of congenital anomaly
* Mechanical ventilator support
* Absence of comorbid disease
* Not having undergone surgery
* No analgesic medication has been administered in the last hour

Exclusion Criteria:

• Infants with diseases such as sepsis that interfere with the application of touch technique

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Score | Data will be collected from 5 minutes before the aspiration up to the 15th minute. Change in this time intervals will be assessed during 15 minutes.
  Pain will be evaluated using the Neonatal Pain Agitation and Sedation Scale (N-PASS).This scale was developed for preterm and term babies. The Turkish validity and reliability study was conducted in 2017. Crying, irritability, behavior-state, facial expression, extremity tone, and vital signs parameters are evaluated in the N-PASS scale. In this scale is evaluated with triple likert type and pain score can be between "0" and "10". Permission was obtained from the authors to use the scale.
Change in Oxygen saturation | Data will be collected from 5 minutes before the aspiration up to the 15th minute. Change in this time intervals will be assessed during 15 minutes.
  Oxygen saturation will be evaluated using the pulse oximeter
Change in Heart rate | Data will be collected from 5 minutes before the aspiration up to the 15th minute. Change in this time intervals will be assessed during 15 minutes.
  Heart rate will be evaluated using the monitor

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Acibadem Health Group Ataşehir Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nist MD, Robinson A, Harrison TM, Pickler RH. An integrative review of clinician-administered comforting touch interventions and acute stress responses of preterm infants. J Pediatr Nurs. 2022 Nov-Dec;67:e113-e122. doi: 10.1016/j.pedn.2022.08.020. Epub 2022 Sep 20. PMID 36137912
- [Background] Dur S, Caglar S, Yildiz NU, Dogan P, Guney Varal I. The effect of Yakson and Gentle Human Touch methods on pain and physiological parameters in preterm infants during heel lancing. Intensive Crit Care Nurs. 2020 Dec;61:102886. doi: 10.1016/j.iccn.2020.102886. Epub 2020 Jun 27. PMID 32601011
- [Background] Im H, Kim E. Effect of Yakson and Gentle Human Touch versus usual care on urine stress hormones and behaviors in preterm infants: a quasi-experimental study. Int J Nurs Stud. 2009 Apr;46(4):450-8. doi: 10.1016/j.ijnurstu.2008.01.009. Epub 2008 Mar 18. PMID 18353332
- [Background] Bahman Bijari B, Iranmanesh S, Eshghi F, Baneshi MR. Gentle Human Touch and Yakson: The Effect on Preterm's Behavioral Reactions. ISRN Nurs. 2012;2012:750363. doi: 10.5402/2012/750363. Epub 2012 Jun 25. PMID 22792482